CLINICAL TRIAL: NCT00560664
Title: Phase 3 Study Comparison of Autologous Chondrocyte Implantation Versus Mosaicoplasty
Brief Title: Comparison of Autologous Chondrocyte Implantation Versus Mosaicoplasty: a Randomized Trial
Acronym: Cartipatch
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB-01-C-01-OT; RB 06.031
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2014-07

CONDITIONS: Knee Chondral or Osteochondral Defect
Keywords: knee; chondral defect; osteochondral defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Autologous chondrocytes transplantation
  Interventions: Procedure: Autologous chondrocytes transplantation
- 2 (Active Comparator): Mosaicoplasty
  Interventions: Procedure: Mosaicoplasty

INTERVENTIONS:
Procedure: Autologous chondrocytes transplantation — Cartilage was harvested, then transferred for cell isolation and culture. Cells are suspended in agarose and transferred to cylindrical molds and surgically implanted 4 weeks later.
  Other Names: Tissue Bank France
  Arms: 1
Procedure: Mosaicoplasty — Osteochondral patch are sampled and then implanted during the same surgical procedure
  Arms: 2

SUMMARY:
Numerous surgical techniques have been developped for the treatment of chondral and osteochondral defects of the knee. Among those techniques autologous chondrocyte transplantation (ACT) was promising but have potential drawbacks. A novel development by TBF is available. The aim of this randomized trial is to compared this new ACT technique to mosaicoplasty. Final outcomes were measured at 2 years using clinical evaluation scoring system (International Knee Documentation Committee), MRI and arthroscopy with biopsy. 64 patients are needed to detect a mean IKDC difference of at least 15 points with 90% power at a 5% alpha level. Twelve surgical centers in France are involved.

ELIGIBILITY:
Inclusion Criteria:

* isolated femoral osteochondral lesion
* aged 18 to 50
* grade 3 or 4 lesion (ICRS) sized 2,5 cm2 to 7,5 cm2.
* IKDC score below 55

Exclusion Criteria:

* pregnancy
* allergy
* arthrosis
* varus or valgus angle greater than 10°
* ACL laxity
* Severe chronic disease
* BMI > 30 Kg/m2
* HIV, B or C Hepatitis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2007-04; Primary Completion 2012-10 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation scoring system | IKDC

SECONDARY OUTCOMES:
MRI | at 2 years
Arthroscopy with biopsy | at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: F DUBRANA, PhD MD, Principal Investigator — University Hospital, Brest
Locations (12):
- France (12):
  - CHU de Lyon, Lyon, Lyon
  - Orthopaedic surgery Departement Brest University Hospital, Brest
  - CHU de Caen, Caen
  - Centre médico chirurgical de Dracy-Le-Fort, Dracy-le-Fort
  - CHU de Grenoble, Grenoble
  - Ch Versailles, Le Chesnay
  - Clinique Chenieux, Limoges
  - CH Nord Mayenne, Mayenne
  - CHU de Nancy, Nancy
  - HIA Bégin, Saint-Mandé
  - CHU de Strasbourg, Strasbourg
  - Clinique du cours Dillon, Toulouse

REFERENCES:
- [Result] Clave A, Potel JF, Servien E, Neyret P, Dubrana F, Stindel E. Third-generation autologous chondrocyte implantation versus mosaicplasty for knee cartilage injury: 2-year randomized trial. J Orthop Res. 2016 Apr;34(4):658-65. doi: 10.1002/jor.23152. Epub 2016 Jan 18. PMID 26742454